CLINICAL TRIAL: NCT05220800
Title: Effects of Intravenous Administered Iron in Non-anemic Iron Deficient Patients With Colorectal Cancer: A Double Blinded Clinical Randomized Trial
Brief Title: Effects of Intravenous Administered Iron in Non-anemic Iron Deficient Patients With Colorectal Cancer
Acronym: NAIDIC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Randers Regional Hospital (Other); Slagelse Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REG-180-2020
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-01

CONDITIONS: Iron-deficiency; Colorectal Cancer
Keywords: surgery; Iron-deficiency; Colorectal cancer; Intravenous iron
MeSH Terms: conditions — Anemia, Iron-Deficiency; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Double-blinded clinical randomized trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Concealement by opaque infusion bags and iv. drips.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron(III)isomaltoside 1000 (Experimental): Weight-dependent one-time dosage of intravenous administration of iron(III)isomaltoside given prior to surgery. Dosage: <50 kg body weight = 500 mg, 50-59 kg body weight = 600 mg, 60-59 kg body weight = 700 mg, 70-79 kg body weight = 800 mg, 80-89 kg body weight = 900 mg, and 90+ kg body weight = 1000 mg.
  Interventions: Drug: Iron(III)isomaltoside
- Placebo (Placebo Comparator): 500 ml isotonic saline infusion fluid
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Iron(III)isomaltoside — Weight-dependent dosage of iron(III)isomaltoside. See group descriptions
  Arms: Iron(III)isomaltoside 1000
Drug: Placebo — Isoton saline infusion
  Arms: Placebo

SUMMARY:
This double-blinded clinical randomized trial with a 1:1 recruitment ratio between placebo and the active group will aim to investigate the effects of intravenously administered iron in non-anemic iron deficient patients on physical capacity, immunological cells and their function prior to surgery. A total of 134 patients with colorectalcancer will be included in the study.

Study outline:

After initial inclusion the patient will undergo baseline testing with cardiopulmonary exercise test (CPET), then followed by an infusion of a weight dependent dosage of iron(III)isomaltoside or placebo. Then at the closest possible time to the surgery the patient will have drawn bloodwork and be re-tested by (CPET). The patient will be followed after surgery with evaluation of several outcomes including quality of recovery and complications. Further, the effects of the intervention on the patients immune function will be evaluated by two different methods: 1) by changes in neutrophil-to-lymphocyte ratio between baseline and preoperative bloodwork and 2) by evaluation mRNA expression in the tumor specimen by the Nanostring pancancer immune panel

DETAILED DESCRIPTION:
Aim The aim is to investigate the effects of intravenously administered iron in non-anemic iron deficient patients on physical capacity, immunological cells and their function prior to surgery.

Study design The study will be performed as a double-blinded clinical randomized trial with a 1:1 recruitment ratio between placebo and the active group. The study will be performed as a multicenter study with inclusion at Department of Surgery, Zealand University Hospital, Departement of Surgery, Slagelse Hospital and Department of Surgery, Regionshospital Randers. The study will need 134 participants, 67 in each arm.

Potential patients will be identified through routine blood samples taken prior to the first consultation. The samples will contain a complete anemia workup and a white blood cell count. The clinical guidelines for identifying and treating anemia in patients with colorectal cancer prior to surgery defines anemia by a hemoglobin ≤ 7 mmol/L for both men and women. Therefore non-anemic patients are defined by a hemoglobin above 7 mmol/L for both men and women in this protocol. Patients, who consents to the study, will immediately after the consultation be randomized and given weight dependent dose of Monofer® (Iron(III)-Isomaltoside) or placebo. On the day prior to surgery (or closest possible time) blood samples similar to the previous samples, will be taken, but with two additional blood samples, which will be stored for later analysis.

At the day of surgery, samples from the invasive front of the removed tumor will be taken and stored for later analysis by the Nanostring PanCancer Immune panel.

The first 20 patients from the Zealand University Hospital and Slagelse hospital will be physical tested by CPET prior to randomization and the day prior to surgery.

All patients will receive the same standardized peri- and postoperative care. All clinical decisions will be at the surgeon's discretion. On the days after surgery until discharge, daily routine blood samples will be taken, including white blood cell count and an assessment of the recovery, through the validated and translated questionnaire Quality of Recovery-15 (QoR-15). Discharge will be handled through standardized discharge criteria. After thirty days after surgery the patient will be contacted by phone for a follow up, concerning complications after discharge and medical records scrutinized for postoperative events.

Randomization and allocation concealment Randomization to the intervention or placebo group will be handled through an online block randomization stratificatied by sex, center of treatment and hemoglobin levels at baseline. Hemoglobin levels at baseline will be divided into four groups: 7.1-8.0, 8.1-9.0, 9.1-10.0 and ≥10.1. Placebo or MonoFer (Iron(III)-Isomaltoside) will be administered through identical opaque bags. Placebo will be an isotonic saline solution. The randomization key will be stored online behind an encryption key (in EasyTrial), which only will be opened after all testing of primary outcomes have been concluded. In order to secure double blinding a specific procedure for administration will be performed outlined in figure 3. When randomization are performed the randomization ID will have a corresponding closed cardboard box with a label with the randomization ID. The box will contain everything needed for concealment, equipment for intravenous administration, isotonic saline solution, and if active also 1000 mg (maximum dosage) MonoFer (Iron(III)-Isomaltoside). The box will be delivered to a clinical nurse which will mix the drug and put it into the opaque bag. A project nurse will secure an intravenous catheter, tape the catheter with opaque tape, put the patients hand through a curtain and leave the room. The clinical nurse will then administer the drug/placebo behind the curtain. The project nurse will do the observation of the patient during the infusion and the clinical nurse will remove the drug/placebo after end infusion. The box will be packed by the Central Pharmacy of Region Zealand and delivered to each site. All clinical nurses will receive training prior to initiation of the study in regards to proper mixing and concealment procedure.

Trial medication, packaging, labeling and administration The trial medication in use for this trial is weight depended MonoFer (Iron(III)isomaltoside 100 mg/ml) versus placebo which is isotonic saline, as an one-time dosage administered intravenously in hospital. The weight depended dosages are as follows: <50 kg bodyweight: 500 mg, 50-59 kg bodyweight: 600 mg, 60-69 kg bodyweight: 700 mg, 70-79 kg bodyweight: 800 mg, 80-89 kg bodyweight: 900 mg, and ≥90 kg bodyweight 1000 mg Monofer. MonoFer needs to be mixed with isotonic saline just prior to administration. Thus, in order to secure proper concealment everything needing for mixing and administration are packed in closed cardboard boxes. The boxes are labelled in concordance with The Rules Governing Medicinal Products in the European Union Directive 2003/94/EC

Each cardboard box will contain 500 ml isotonic saline infusion fluid, a drop line and an opaque bag which will cover both the line and the fluid, labeling for the opaque bag, and a standard operating procedure document detailing handling and allocation concealment procedure (appendix II: Håndtering af forsøgsmedicin). If allocated to the active group the box will also contain 10ml MonoFer 100mg/ml.

If the administration are interrupted before the full dosage are administered the actual dosage given are noted by the clinical nurse and passed on to the project nurse which will secure the registration without deblinding the patient or research staff. Otherwise the full dosage of 500 ml will be recorded.

The infusion will be stopped if the patient experiences any adverse effects during the infusion. A particular reaction called a 'Fishbane reaction' in which the patient develops reddening of the skin, especially in the face, and truncal myalgia, but without any other symptoms of an allergic reaction will not be cause termination of the infusion. The Fishbane reaction is always selflimitating and is not associated with respiratory stridor, edema, hypotension or tachycardia. In case of a Fishbane reaction the infusion is stopped until the symptoms have dissipated, then the infusion is restarted, but with double the infusion time. If the Fishbane reaction reoccurs the infusion is terminated and dosage given registered.

Definition of per protocol Patients are considered per protocol if the patient received full dosage of placebo or MonoFer, and underwent surgery for a malignant tumor.

ELIGIBILITY:
Inclusion Criteria:

* Planned for curative intended elective colon or rectum cancer surgery
* UICC stage I-III (at diagnosis)
* Hemoglobin > 7.0 mmol/L
* Serum ferritin <101 microgram/L or transferrin saturation <21%

Exclusion Criteria:

* Chronic kidney failure with need for dialysis
* Metachronous diagnosed cancer
* Unable to speak or understand Danish
* Cognitive impairment e.g. moderate to severe dementia
* Concurrent severe active bacterial infection
* Known allergy for Iron(III)isomaltoside
* Contraindications for intravenous iron (Pofryria, livercirrosis, active hepatitis, transaminases three times the upper limit, hemosiderosis and hemochromatosis)
* Withdrawal of informed consent
* Neoadjuvant chemo or radiation therapy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in oxygen uptake at the anaerobic threshold | at baseline and 1-4 days before surgery
  Change in oxygen uptake at the anaerobic threshold measured by cardiopulmonary exercise test before infusion and the days before surgery
Change in neutrophile to lymphocyte ratio (NLR) | at baseline and 1-4 days before surgery
  Change in neutrophile to lymphocyte ratio (NLR) between baseline bloodwork and prior to surgery.
Changes in T-cell function - mRNA expression analysis | 1 day after surgery
  Nanostring pancancer immune analysis of tumor samples

SECONDARY OUTCOMES:
Quality of Recovery 15 (QoR-15) | Up to 7 days after surgery
  Questionaire Quality of Recovery 15 (QoR-15). Scale of 15 questions regarding surgical recovery. Each item with a maximum score of 10 and minimum of 0. Total maximum score 150. Lowest 0. The higher score the better recovery
Complications | 30-days after surgery
  Postoperative complications graded by the Clavien-Dindo classification and the comprehensive complication index
Days alive and out of hospital - 30 | 30 days after surgery
  Days alive and out of hospital 30 days after surgery
1 year cancer free survival | 1 year after surgery
  1 year cancer free survival. Either death or recurrence
5 year cancer free survival | 5 years after surgery
  5 year cancer free survival. Either death or recurrence

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Zealand University Hospital, Køge, Danmark
  - Slagelse Hospital, Slagelse, Danmark
  - Regionshospitalet Randers, Randers